CLINICAL TRIAL: NCT00788866
Title: Impact of Maternal Pomegranate Juice on Brain Injury in Infants With Intrauterine Growth Restriction (IUGR)
Acronym: POM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: POM Wonderful LLC (Industry); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Methodius Tuuli, MD, MPH, Assistant Professor, Washington University Early Recognition Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: Pomegranate-1
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Intrauterine Growth Restriction
Keywords: Neuroprotection; Antioxidants; Neonatal brain injury; Pomegranate juice
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate juice (Experimental): This arm with receive 8oz of pomegranate juice per day.
  Interventions: Dietary Supplement: Pomegranate Juice
- Placebo (Placebo Comparator): This group will take 8oz of placebo juice that lacks pomegranate daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice — 8 oz of pomegranate juice daily vs placebo juice identical in all respects except pomegranate
  Arms: Pomegranate juice
Dietary Supplement: Placebo — Juice that matches the makeup of pomegranate in regards to sugar, vitamin C, etc. The only difference is that it lacks pomegranate juice.
  Arms: Placebo

SUMMARY:
Infants with intrauterine growth restriction are known to be at increased risk for long term neurodevelopmental delay into adulthood. The main mechanism for this is likely decreased blood flow to the brain secondary to altered placental blood flow. Antioxidants may serve to protect the developing brain from this process. Animal studies have shown that pomegranate juice protects the fetal brain from injury in a model of stroke. This clinical trial is intended to evaluate if giving mothers pomegranate juice during the last several weeks of pregnancy can help protect intrauterine growth restricted babies' brains.

DETAILED DESCRIPTION:
This study is divided into two separate phases.

Phase I evaluated if the antioxidants produced from pomegranate juice cross the placenta in normal healthy pregnancies. Twenty women were enrolled, 10 who will take 8 oz of pomegranate juice daily and then 10 others who will take 8 oz of placebo juice without pomegranate daily. Blood samples were first collected from the woman at the time enrollment and then from both the woman and the cord blood at the time of delivery. These blood samples were analyzed to measure the levels of antioxidant metabolites from the pomegranate juice. This phase was deigned to confirm placental transfer of antioxidant pomegranate metabolites. The results confirmed placenta transfer of pomegranate metabolites. Further, placental tissues from 12 patients (4 in the pomegranate group and 8 in the control group) were collected for analysis of oxidative stress. The preliminary in vivo results were extended to oxidative stress and cell death assays in vitro. Placental explants and cultured primary human trophoblasts were exposed to pomegranate juice or glucose (control) under defined oxygen tensions and chemical stimuli. We found decreased oxidative stress in term human placentas from women who labored after prenatal ingestion of pomegranate juice compared with apple juice as control. Moreover, pomegranate juice reduced in vitro oxidative stress, apoptosis, and global cell death in term villous explants and primary trophoblast cultures exposed to hypoxia, the hypoxia mimetic cobalt chloride, and the kinase inhibitor staurosporine. Punicalagin, but not ellagic acid, both prominent polyphenols in pomegranate juice, reduced oxidative stress and stimulus-induced apoptosis in cultured syncytiotrophoblasts.

Phase II focuses on pregnancies with intrauterine growth restriction. If they meet entry criteria, then woman will be enrolled and randomized into 1 of 2 groups.

Treatment group: Expecting mothers in this group will start a daily regimen of 8 oz glass of pomegranate juice. They will keep a daily diary documenting their compliance. They will continue this daily intake up until delivery of their infant.

Placebo group: These women will start a daily regimen of an 8 oz of pomegranate free juice placebo that matches taste, calories, and appearance to regular pomegranate juice but lacks polyphenols. They will also keep a diary of daily intake to help ensure compliance similar to the treatment group. They too will continue to take the placebos up until the time they deliver.

Both groups: All women will be followed up on a weekly basis to assess compliance. A detailed diet history will be collected from the women at the time of enrollment, midway through the 3rd trimester and at the time of delivery. Furthermore, all women will have a detailed social history collected at the time of enrollment. Upon delivery, cord blood will be collected and sent for ellagic acid, a polyphenic component. All placental material will be sent for formal pathological exam and analyzed for markers of placental injury.

If clinically stable, the infants will receive MRI evaluations to evaluate for possible brain injury.

ELIGIBILITY:
Phase I:

Inclusion Criteria:

* Healthy expecting mothers two weeks from their expected due dates
* No evidence of IUGR
* No evidence of fetal problems

Phase II:

Inclusion Criteria:

1. Expecting mother with a fetal diagnosis of intrauterine growth restriction (IUGR) defined by estimated fetal weight <10th percentile for gestational age
2. 24 - 34 weeks gestation

Exclusion Criteria:

1. Major congenital abnormalities
2. Known fetal chromosomal disorder
3. Maternal illicit drug use
4. Maternal IV and Hepatitis C infection
5. Premature rupture of membranes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
CNS injury at term by MR Imaging | 36 - 41 weeks (post delivery)
  1. Qualitative MRI injury- white matter injury (WMI) and gray matter injury (GMI)
  2. Brain Metrics on MR imaging
  3. Diffusion- apparent diffusion coefficient (ADC) and fractional anisotropy (FA)
  4. Spectroscopy- lactate and NAA levels in the basal ganglia
  5. Advanced MRI development indices - brain volumes, surface based morphology (SBM, folding indices)

SECONDARY OUTCOMES:
Placental morphology: weight and size | At birth
Gestational age at delivery | At birth
Birth weight | At birth
Ellagic acid levels from cord blood | To discharge
Dubowitz neurologic exam at term | To discharge
Time to full oral feeds | To discharge
ROP | To discharge
NEC | To discharge
Length of ventilatory support | To discharge
Time to discharge | To discharge
Placental micrography: number of villi, vasculature, collagen content | At birth
Placental immunohistochemistry: proliferation, apoptosis and differentiation | At birth
Placental: immunoassays: HSP90, lipid hydroperoxide, nitrotyrosine assay, paraoxonase 1 expression, superoxide dismutases | At birth
Placental RNA microarray | At birth
Umbilical cord gases | At birth
Pregnancy complications: preeclampsia | At birth
Neonatal wellbeing: APGAR scores, need for resuscitation | At birth

OTHER OUTCOMES:
Maternal compliance | To delivery
  1. Daily dietary report
  2. Increase in polyphenol levels
Analysis both by 'intention to treat' and 'as treated' | To discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nelson, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- St Louis Children's Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Matthews LG, Smyser CD, Cherkerzian S, Alexopoulos D, Kenley J, Tuuli MG, Nelson DM, Inder TE. Maternal pomegranate juice intake and brain structure and function in infants with intrauterine growth restriction: A randomized controlled pilot study. PLoS One. 2019 Aug 21;14(8):e0219596. doi: 10.1371/journal.pone.0219596. eCollection 2019. PMID 31433809